CLINICAL TRIAL: NCT00883974
Title: Early Sensitivity Training for Parents of Preterm Infants: Impact on the Developing Brain
Brief Title: Sensitivity Training For Parents of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: The Financial Markets Foundation for Children (Other)
Responsible Party: Jeannette Milgrom, University of Melbourne & Austin Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Preterm Sensitivity Training
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Development; Preterm Birth
Keywords: preterm bith; neurodevelopment; sensitivity training; magnetic resonance imaging (MRI); Infant neurodevelopment following preterm birth
MeSH Terms: conditions — Premature Birth | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Sensitivity Training
- 2 (No Intervention): Standard Neonatal Intensive Care Unit (NICU) procedures for the care of pre-term infants

INTERVENTIONS:
Behavioral: Sensitivity Training — The parent sensitivity training program was delivered in NICU (9 sessions) with a home-booster session. Therapists worked with parents following a manualized protocol. Targets of intervention included: recognizing signs of infant stress, "shut-down" mechanisms, alert-available behavior, motor behaviors, facial expressions,posture/muscle tone; graded stimulation; how to optimize interactions; touch, movement and massage; "kangaroo care" (nesting infants skin-to-skin against their mother); vocal, visual and multi-sensory stimulation; normalizing parental feelings; challenging dysfunctional thinking, and diary keeping.
  Arms: 1

SUMMARY:
Immediately following birth, preterm infants face a period of stressful environmental inputs, which may have negative consequences on early brain development and subsequent neurobehavioral outcomes. This study aimed to assess the effectiveness of training parents in reducing stressful experiences early in life. The investigators hypothesized that this intervention would insulate preterm infants from the harmful effects of acute and chronic stress, which in turn would result in enhanced brain development. The primary aim of the current study was to investigate if this intervention was associated with improved brain development measured by magnetic resonance imaging (MRI) at term-equivalent age. A secondary aim was to assess some possible short-term medical benefits.

DETAILED DESCRIPTION:
A randomized controlled trial of a parental sensitivity training program involving 45 women with infants born < 30 weeks gestational age. The intervention consisted of 10 individual sessions in the Neonatal Intensive Care Unit (NICU). Post-intervention, at term-equivalent age (40 weeks postmenstrual age), magnetic resonance (MR) imaging was performed to evaluate brain structure and development. Quantitative volumetric techniques were used to estimate overall and regional brain volumes for different tissue types including cerebrospinal fluid (CSF), cortical grey matter (CGM), deep nuclear grey matter (DNGM), unmyelinated white matter (UWM) and myelinated white matter (MWM). Diffusion tensor imaging (DTI) was used to evaluate the integrity and maturation of white matter by apparent diffusion coefficient (ADC) and fractional anisotropy (FA).

ELIGIBILITY:
Inclusion Criteria:

* > 30 weeks gestation

Exclusion Criteria:

* insufficient English
* congenital abnormality
* triplets and higher multiple births
* residence > 100 km from study site

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging | Preterm infants at full-term equivalent age (40 weeks post-menstrual age)

SECONDARY OUTCOMES:
Short-term medical stability | Birth to full-term eqivalent age (40 weeks post-menstrual age)

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Milgrom, PhD, Principal Investigator — University of Melbourne/Austin Health
Locations (2):
- Australia (2):
  - Austin Health, Melbourne, Victoria
  - Jeannette Milgrom, Melbourne, Victoria

REFERENCES:
- [Derived] Milgrom J, Newnham C, Anderson PJ, Doyle LW, Gemmill AW, Lee K, Hunt RW, Bear M, Inder T. Early sensitivity training for parents of preterm infants: impact on the developing brain. Pediatr Res. 2010 Mar;67(3):330-5. doi: 10.1203/PDR.0b013e3181cb8e2f. PMID 19952869